CLINICAL TRIAL: NCT03687775
Title: Intraoperative Stability Assessment of the First Carpometacarpal Joint
Brief Title: CMC I Stability Intraoperative
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: DSG-Stabi
Record Dates: First submitted 2018-09-12; First posted 2018-09-27 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Osteoarthritis Thumb; Arthrosis of First Carpometacarpal Joint; Joint Instability
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DSG-Stabi: The group consists of patients with primary trapeziometacarpal osteoarthritis and an indication for trapeziectomy alone or in combination with the resection-suspension-interposition arthroplasty.
  Interventions: Other: Stability assessment

INTERVENTIONS:
Other: Stability assessment — Qualitative and quantitative stability assessment

SUMMARY:
The goal of the current study is to objectively measure intraoperative the initial thumb stability after trapezium removal when performing trapeziectomy, alone or in combination with suspension and tendon interposition and to evaluate if there are differences in the stability between the patients and with the different surgical steps. Additionally, the subjective stability rating of the surgeon will be compared with the objective measures and if there is a correlation between clinical/patient-related parameters and the measured intraoperative stability.

DETAILED DESCRIPTION:
Osteoarthritis of the first carpometacarpal joint (CMC I OA) treatment strategies typically focus on pain relief and restoring motion and function. Besides different other treatment modalities, such as trapeziectomy (removal of the trapezium bone) alone, the resection-suspension-interposition arthroplasty (after trapezium resection additional stabilisation with a tendon strip) (LRTI) are the most popular interventions. When performing trapeziectomy, alone or in combination with suspension and tendon interposition, the surgeon perceives individual differences in joint stability. However, there are no quantitative data available on the stability of the CMC I joint after trapeziectomy. Furthermore, the relative contribution of the different surgical steps to the stability of the joint is unknown. The goal of the current study is to objectively measure intraoperative thumb stability and evaluate if there are differences in the stability between the patients and with the different surgical steps. Additionally, the subjective stability rating of the surgeon will be compared with the objective measures. Additionally, the subjective stability rating of the surgeon will be compared with the objective measures and if there is a correlation between clinical/patient-related parameters and the measured intraoperative stability.

Procedure 1: Patient enrollment

During the preoperative consultation, the surgeon identifies patients which meet the inclusion criteria. Before any study specific examinations are performed, the patient has to give written informed consent to participate in the study according to the clinical investigation protocol. Patients will have enough time to decide for or against participation until before the surgery (usually one-six weeks after the consultation).

Baseline data:

After inclusion in the study, documented by patient informed consent, the following data will be collected:

* Z-deformity will be measured with a goniometer.
* Grip strength of the affected hand will be measured with the help of a Jamar dynamometer and key pinch will be measured using a pinch gauge. Both measurements are performed three times. For each of these, the average of the three measurements is taken. The standardized testing position as recommended by the American Society of Hand Therapists will be used.
* The ability to oppose the thumb will be quantified using the Kapandji index.
* Joint laxity will be quantified using the Beighton Hypermobility Score.
* X-rays will be rated for the stage of OA according to the criteria described by Eaton & Littler.

Furthermore, the participant answers questions about his/her hand usage in daily life, pain and completes the brief Michigan Hand Outcomes Questionnaire.

Procedure 2: Surgery

Stability Assessment:

After trapeziectomy according to the standard surgical procedure, the surgeon subjectively rates the CMC I joint stability (stable, somewhat stable and instable) by displacing the thumb proximally. The objective stability measurement is performed after the subjective assessment: The hand is standardized positioned in a pinch grip position. A standard reposition forceps is attached to the base of the first metacarpal bone. Next, the reposition forceps is connected to the force sensor and the thumb ray displaced by 10 mm towards the scaphoid with a guide. While the counteracting forces are measured with a force sensor. This procedure is applied by the surgeon after every step of the LRTI surgery:

1. Trapeziectomy
2. Suspension
3. Interposition
4. Closing of the joint capsule

The measurement is repeated three times for every step. A high value indicates high stability. For blinding purposes, the surgeon will not see the measurement results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with primary trapeziometacarpal osteoarthritis in the thumb and indication for LRTI surgery
* Indication for Trapeziectomy alone
* Informed Consent as documented by signature
* Patient aged 18 years and over

Exclusion Criteria:

* Previous surgeries of the affected CMC I joint
* Inflammatory disease (e.g. rheumatoid arthritis)
* Tumour / malignoma
* German language barrier to complete the questionnaire
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* Legal incompetence
* Indication for pyrocarbon implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with CMC I joint osteoarthritis and an indication for LRTI. In the Schulthess Klinik, around 150 interventions of resection of the trapezium with LRTI are performed per year. Therefore many patients are available.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Primary thumb stability in newton measured with DaSta | intraoperative period
  Objective primary thumb stability after trapeziectomy measured in newton (kg*m/s2) with the DaSta measurement system

SECONDARY OUTCOMES:
Thumb stability in newton measured with DaSta after suspension, interposition and joint capsule closure | intraoperative period
  Objective thumb stability measured in newton (kg*m/s2) with the DaSta measurement system after:
  * Suspension
  * Interposition
  * Closing of the joint capsule
Qualitative primary thumb stability in 3 point rating scale | intraoperative period
  Surgeon rates qualitatively the primary thumb stability (stable, somewhat stable and instable) after trapeziectomy by displacing the thumb in proximal direction.
Correlation and relationship between all patient-related and clinical parameters with the measured stability | Pre Operation
  Correlation and relationship between all patient-related and clinical parameters with the measured stability.
  Clinical parameters:
  * Socio-demographic data (includes: BMI, dominant hand)
  * Objective functional parameters (Z- deformity, key pinch strength, grip strength, Kapandji index, Beighton Hypermobility Score, Eaton Stage of thumb carpometacarpal joint osteoarthritis)
  * Subjective functional parameters (brief Michigan Hand Questionnaire, pain level by numeric rating scale, hand use in daily life)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B. Herren, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No